CLINICAL TRIAL: NCT01276405
Title: The Efficacy of Adjuvant Chemotherapy With Capecitabine (Xeloda) Monotherapy in Patients With Colon Cancer Stage III (Duke C) Considering the Histopathology of the Tumour (AXEL)
Brief Title: An Observational Study of Xeloda (Capecitabine) Monotherapy in Patients With Colorectal Cancer (AXEL)
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25174
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate Xeloda (capecitabine) monotherapy on the effect of disease-free survival in patients with colon cancer stage III (Duke C) after surgical resection. Data will be collected for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, over the age of 18 years
* Presence of colon adenocarcinoma
* Surgical resection for colon cancer stage III (Duke C)
* Prior adjuvant therapy with Xeloda monotherapy

Exclusion Criteria:

* Contraindications for Xeloda

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer stage III (Duke C) on Xeloda monotherapy
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2010-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

SECONDARY OUTCOMES:
Safety (Incidence of adverse events) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bucharest, Romania